CLINICAL TRIAL: NCT03219008
Title: Multi-dimensional Diagnosis,Individualized Therapy,and Management Technique for Major Depressive Disorder:Based on Clinical and Pathological Characteristics
Acronym: STEP-MDD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Chinese Academy of Sciences (Other Government); Shanxi Medical University (Other); Central South University (Other); Second Military Medical University (Other); Peking University Sixth Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Kunming Medical University (Other); Air Force Military Medical University, China (Other); Zhejiang University (Other); Wuhan Mental Health Centre (Other); Corning Hospital, Shenzhen City (Unknown); the First Specialized Subject Hospital of Harbin (Unknown); Renmin Hospital of Wuhan University (Other); Seventh People's Hospital of Hangzhou (Other); Shandong Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016YFC1307100
Record Dates: First submitted 2017-05-07; First posted 2017-07-17 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-05

CONDITIONS: Depressive Disorder
Keywords: depressive disorder; multi-dimensional diagnosis technique; individualized therapy; management technique; e-MBC; MBC
MeSH Terms: conditions — Depressive Disorder | interventions — Fluoxetine; Bupropion; Fluvoxamine; Lithium; Physical Therapy Modalities; Mirtazapine; Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: Part 2: all patients before receiving any medicine treatment are divided into four groups which adopt different therapy strategies :treatment with fluvoxamine, fluoxetine, mirtazapine and treatment as usual(TAU).Meanwhile，patients with different subtypes of depressive disorder were randomly assigned to different therapy groups.Each therapy groups contains 50 participants.Therefore, the total sample size is 50*12+200=800.
  Part3:To find out efficiency of different kinds of therapy strategies.p=60%, error=5%,a-0.05,the amount of samples nearly is:867,considering the nearly 30% expulsion rate, the final total sample size is 867+260=1127.Therefore,sample size in each group is nearly 376.
  Part4:p=60%,error=0.05, a=0.05, exculsion rate=30%,N=867+260=1127.the amount of samples of each group is 1127/3=nearly 400.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients with depressive disorder were randomly assigned to different therapy groups or TAU therapy group based on different depressive disorders subtypes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Depression/underload 1 (Experimental): This group would be treated with fluoxetine from the minimum dosage.
  Interventions: Drug: Fluoxetine
- Depression/underload 2 (Experimental): This group would be treated with fluoxetine combined with cognitive behavior treatment
  Interventions: Combination Product: fluoxetine + cognitive-behavioral treatment（CBT）
- Depression/underload 3 (Experimental): This group would be treated with fluoxetine and amfebutamone from the minimum dosage.
  Interventions: Drug: fluoxetine + Amfebutamone
- Depression/underload 4 (Experimental): This group would be treated with fluoxetine + physical treatment to help to cure depressive disorder.
  Interventions: Combination Product: physical treatment+fluoxetine+amfebutamone
- Atypical 1 (Experimental): This group would be treated with fluvoxamine from the minimum dosage.
  Interventions: Drug: Fluvoxamine
- Atypical 2 (Experimental): This group would be treated with fluoxetine + cognitive behavior treatment
  Interventions: Combination Product: Cognitive behavior treatment +fluvoxamine
- Atypical 3 (Experimental): This group would be treated with fluvoxamine + lithium from the minimum dosage.
  Interventions: Drug: Lithium+fluvoxamine
- Atypical 4 (Experimental): This group would be treated with fluvoxamine + lithium + physical treatment
  Interventions: Combination Product: fluvoxamine + lithium + physical therapy
- Anxiety/somatization 1 (Experimental): This group would be treated with mirtazapine/selective serotonin-norepinephrine reuptake inhibitors（SNRIs） from the minimum dosage.
  Interventions: Drug: Mirtazapine/SNRIs
- Anxiety/somatization 2 (Experimental): This group would be treated with mirtazapine/SNRIs + cognitive behavior treatment.
  Interventions: Combination Product: mirtazapine+ Cognitive behavior treatment
- Anxiety/somatization 3 (Experimental): This group would be treated with mirtazapine + SNRIs from the minimum dosage.
  Interventions: Drug: mirtazapine + SNRIs
- Anxiety/somatization 4 (Experimental): This group would be treated with mirtazapine + SNRIs + physical treatment.
  Interventions: Combination Product: mirtazapine + SNRIs + physical therapy
- treatment as usual(TAU) (Experimental): The investigators recommend therapy strategies according to accessible methods.
  Interventions: Other: TAU(treat as usual)

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine is one kind of selective serotonin reuptake inhibitor(SSRIs), whose effect is much better than other non-underload subtypes compared with underload subtypes.So patients would be treated with fluoxetine only.
  Arms: Depression/underload 1
Combination Product: fluoxetine + cognitive-behavioral treatment（CBT） — the investigators would recommend fluoxetine to help to cure depressive disorder.And CBT is a very effective way for patients to alleviate or relieve clinical symptoms during episode stage.
  Arms: Depression/underload 2
Drug: fluoxetine + Amfebutamone — Amfebutamone is one kind of SNRIs, and it shows much better therapy effect on patients with exhaustion /dizziness.So the investigators recommend these two drugs to help to cure patients with depressive disorder.
  Arms: Depression/underload 3
Combination Product: physical treatment+fluoxetine+amfebutamone — the investigators recommend drug(fluoxetine and amfebutamone) and physical treatment as intervention.
  Arms: Depression/underload 4
Drug: Fluvoxamine — Fluvoxamine could inhibit CYP1A2 and CYP2C19 and affect the metabolism of melatonin, and help to release symptoms of depressive disorder with sleep problems.
  Arms: Atypical 1
Drug: Lithium+fluvoxamine — the investigators recommend lithium as a mood stabilizer and use fluvoxamine to affect the level of melatonin.
  Arms: Atypical 3
Combination Product: fluvoxamine + lithium + physical therapy — the investigators recommend depressants and mood stabilizers as well as physical therapy to help to cure depressive disorder.
  Arms: Atypical 4
Combination Product: Cognitive behavior treatment +fluvoxamine — the investigators recommend behavioral therapy as well as drugs.
  Arms: Atypical 2
Drug: Mirtazapine/SNRIs — Mirtazapine is one kind of antagonist of a2 adrenergic receptors and could block 5-hydroxytryptamine2 and 5-hydroxytryptamine3,help to release symptoms like anxiety or somatization.Besides, SNRIs could also make similar effect on patients.Therefore, the investigators recommend mirtazapine/SNRIs to treat patients with depressive disorder.
  Arms: Anxiety/somatization 1
Combination Product: mirtazapine+ Cognitive behavior treatment — the investigators recommend CBT and mirtazapine as interventions.The dosage and frequency would depend on patients' severity of symptoms .
  Arms: Anxiety/somatization 2
Drug: mirtazapine + SNRIs — the investigator recommend mirtazapine and SNRIs to treat patients with major depressive disorder.
  Arms: Anxiety/somatization 3
Combination Product: mirtazapine + SNRIs + physical therapy — the investigators would manage to use drugs and physical treatment to help to release the symptoms of depressive disorder.
  Arms: Anxiety/somatization 4
Other: TAU(treat as usual) — patients in this group would receive therapy strategies according to their symptoms and preference.
  Arms: treatment as usual(TAU)

SUMMARY:
Major Depressive Disorder is one of the most common mental diseases,which increases health-care costs and the financial burden to families and societies. Considering its complex clinical symptoms and diversity of comorbidity, depressive disorder's recognition，diagnosis，and antihistone are based on symptomatology,which is lack of multidimensional diagnosis technique based on clinical pathological characteristics,as well as lack of individualized therapy strategy based on quantified evaluation. Besides, other physical diseases，such as nervous system diseases, cardiovascular diseases，endocrine diseases, have the high comorbidity of depressive disorder. However，there is no precise diagnosis technique or standardized therapy strategy. With all those taken into consideration,our study is aimed to adopt E-mental health and m-Health to explore multi-dimensional diagnosis, individualized therapy and management technique based on molecular biology,nerve electrophysiology，and neuroimaging technology etc.

DETAILED DESCRIPTION:
Four parts included in our study:

Part 1:The research, development and verification of indicators based on biomarkers and clinical characteristics to guide the diagnosis and treatment of depressive disorders

1. to screen biomarkers, to explore its pathophysiology, and to analyze the correlation between clinical subtypes/characteristics and biomarkers.
2. To differentiate the subtypes of depressive disorder（depression/underload, atypical, anxiety/somatization) based on clinical symptoms and clinical assessement.
3. To establish personalized therapy strategies,and to explore tool kits for diagnosis and treatment based on biomarkers and clinical characteristics.
4. to choose appropriate indicators to monitor therapy and side effect by collecting and analyzing blood/imaging/neuropsychological data.

Part 2: The development,transition and application of hierarchical model diagnostic technique for physical diseases combined with depressive disorder.

1. to recruit patients with physical diseases combined with depressive disorder, and explore potential biomarkers.
2. To chose appropriate therapy strategies based on measurement based care（MBC）, providing hierarchical model diagnostic technique for patients.
3. To weigh therapy efficiency and adverse effect among different medicine therapy groups.

Part3: The development and application of comprehensive prevention， diagnosis,and intervention model of depressive disorder.

1. To explore and establish online screening and assistant diagnosis system for patients with depressive disorder.
2. research ,development and application of intelligent e-MBC. Part 4: The development,transition and application of e-MBC sharing platform.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years;
* clinical diagnosis of major depressive disorder;
* 17-Hamilton Depression Scale>20;
* 14-Hamilton Anxiety Scale score<7;
* outpatient treatment;
* first episode;
* medication-naive;

Exclusion Criteria:

* clinical diagnosis of schizophrenia, schizoaffective disorder;
* any prescription or psychotropic medications in the past 4 week;
* serious medical or neurological illness;
* current pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in levels of microRNA，apolipoproteins, meta ion (Composite measure) | at 2,4,6,8,12 week.
  The potential biomarkers in our study include microRNA,apolipoproteins,metallic ion etc.We use quantitative analysis technique to test miRNA,proteins and metallic ion by patients' blood and urines before interventions and after interventions.

SECONDARY OUTCOMES:
Hamilton Depression Scale(HADA) scores,reductive ratio | at 0,2,4,6,8,12 week.
  HADA,created by Hamilton in 1960,is one of the most common questionnaires to evaluate the severity of depression and the efficiency of medicine. we adopt the Hamilton Depression Scale(HADA)to evaluate different medicines efficiency by analyzing reductive ratio.The investigators record the total scores of HADA at baseline and 2,4,6,8,12 week.
Patient health questionnaire(PHQ-9):the clinical remission ratio | change from baseline PHQ-9 total scores at 2,4,6,8,12 week
  PHQ-9 is a self-report scale composed of 9 items to evaluate the state of depression.The investigators in our study record the total scores of PHQ-9 at 0,2,4,6,8,12 week to analyze the clinical remission ratio.
life event scale(LES) | at baseline
  LES is one of the common questionnaires to evaluate individual's mental and stress stimulation in daily life.The investigators record the total scores of LES at baseline.
social support scale(SSS) | at baseline
  SSS is one of the common questionnaires to evaluate individual's social support and social relationship network to explore the correlation between social support and mental health. the investigators in our study record the total scores of SSS at baseline.
dysfunctional attitudes scales(DAS) | at baseline
  The DAS is a self-report scale composed of 40 items to assess typical, stable depressogenic attitudes or schemas that make individuals vulnerable to depression. The investigators in our study record the total scores od DAS at baseline.
the gray matter volume, | change from baseline neuroimaging data at 2,4,6,8,12 week
  The investigators in our study use voxel-based morphometry (VBM8)to record the gray matter volume.
fractional amplitudes of low-frequency fluctuation(fLAFF) | change from baseline neuroimaging data at 2,4,6,8,12 week
  The investigators in our study use region-of-interest(ROI)to record fLAFF.
Neuroelectrophysiological examination: electroencephalogram(EEG) | at baseline
  EEG is used to record individual's brain activity. The investigators in our study record individual's brain wave.
Neuroelectrophysiological examination:electrocardiograph(ECG) | at baseline.
  ECG is used to record the individual's cardiac cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- ShanghaiMHC, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
To share raw data via the network platform named Clinical Trial Management Public Platform within 1year after the trial finished. And the platform website address is http://www.medresman.org

REFERENCES:
- [Derived] Liu H, Wu X, Wang Y, Liu X, Peng D, Wu Y, Chen J, Su Y, Xu J, Ma X, Li Y, Shi J, Yang X, Rong H, Forti MD, Fang Y. TNF-alpha, IL-6 and hsCRP in patients with melancholic, atypical and anxious depression: an antibody array analysis related to somatic symptoms. Gen Psychiatr. 2022 Sep 8;35(4):e100844. doi: 10.1136/gpsych-2022-100844. eCollection 2022. PMID 36189181
- [Derived] Wang Y, Liu X, Peng D, Wu Y, Su Y, Xu J, Ma X, Li Y, Shi J, Cheng X, Rong H, Fang Y. A Preliminary Study of Different Treatment Strategies for Anxious Depression. Neuropsychiatr Dis Treat. 2022 Jan 4;18:11-18. doi: 10.2147/NDT.S320091. eCollection 2022. PMID 35018097
- [Derived] Liu X, Wang Y, Peng D, Zhang H, Zheng Y, Wu Y, Su YA, Liu M, Ma X, Li Y, Shi J, Cheng X, Rong H, Fang Y. The Developmental and Translational Study on Biomarkers and Clinical Characteristics-based Diagnostic and Therapeutic Identification of Major Depressive Disorder: Study Protocol for a Multicenter Randomized Controlled Trial in China. Neuropsychiatr Dis Treat. 2020 Oct 9;16:2343-2351. doi: 10.2147/NDT.S271842. eCollection 2020. PMID 33116533